CLINICAL TRIAL: NCT02526836
Title: Complete Mesocolic Excision (CME) With Central Supplying Vessel Ligation (CVL) Compared With Conventional Surgery for Colon Cancer: a Double-blinded Randomized Study
Brief Title: Complete Mesocolic Excision With Central Vessel Ligation Compared With Conventional Surgery for Colon Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelkhalek, Assistant Lecturer of Surgical Oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Complete Mesocolic Excision
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2017-11

CONDITIONS: Colon Cancer
Keywords: colon cancer mesocolic excision central ligation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison group (Other): including the number of cases with complete data who underwent surgery using the conventional method.
  Conventional surgery
  Interventions: Procedure: Conventional Surgery
- Intervention group (Active Comparator): including a convenient sample of about 20 patients which is expected to be recruited, for whom Complete Mesocolic Excision (CME) and Central Vascular Ligation (CVL) will be done.
  Complete mesocolic excision with central vascular ligation
  Interventions: Procedure: Complete mesocolic excision with central vascular ligation

INTERVENTIONS:
Procedure: Conventional Surgery — removal of the tumor with no ligation of the vessel centrally or removal of the whole mesocolon
  Arms: Comparison group
Procedure: Complete mesocolic excision with central vascular ligation — excision of the whole mesocolon plus ligation of the supplying blood vessel centrally
  Arms: Intervention group

SUMMARY:
The aim of this study is to compare between complete mesocolic excision with central vascular ligation and conventional surgery of colon cancer regarding number of harvested lymph nodes, surgical outcome and complications.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common human malignant epithelial tumor and still represents the second cause of cancer death in the United States and Europe.

Over the past few decades, there have been significant improvements in the treatment of patients with colonic and rectal cancers. In rectal cancer, the role of earlier diagnosis, improved preoperative staging, neoadjuvant therapy and total mesorectal excision have improved outcomes from oncological and patient recovery perspectives. Of these, arguably the most important for the surgeon was the advent of Total Mesorectal Excision (TME).

Current thinking is that colonic tumors spread via hematogenous, lymphatic, and possibly perineural routes, with the lymphatics anatomically following the arterial supply. Current practice is to excise a proportion of the draining lymphatic bed to accurately stage the cancer and also clear possible lymphatic metastases.

Recently, significant debate has centered on the degree of lymphatic clearance required; several reports have demonstrated improved oncologic outcomes with wider lymphovascular resections compared with current standard practice. Whether these improved outcomes are secondary to improved lymph node yield or an alternative technical effect has not yet been ascertained.

In analogy to total mesorectal excision (TME) for rectal cancer complete mesocolic excision was recently introduced for curative treatment of colon cancer. Like TME, CME aims at complete en bloc clearance of the lymphatic drainage of the tumor enveloped in intact fascias of embryologic origin.

Based on total mesorectal excision experience, further investigations of the importance of complete mesocolic excision and central vascular ligation surgery for colonic cancer were done by comparing a series of complete mesocolic excision and central vascular ligation specimens from Erlangen, Germany to standard excisions from Leeds, United Kingdom. Lymph node yields, tissue morphometry, and grading the plane of surgery were used to investigate differences between the techniques that could potentially explain the relative differences in survival.

The group from Erlangen in Germany have advocated for CME in conjunction with central vascular ligation for colon cancer. Complete mesocolic excision is reported to differ from traditional colon cancer surgery by achieving a far more radical excision of the lymphovascular pedicle and mesocolon. In addition, the complete mesocolic excision technique promotes resection of the specimen with an intact visceral peritoneum together with proximal and distal resection margins of at least 10 cm. Arterial supply to the affected segment of bowel is taken at its origin from the superior mesenteric artery (right and transverse colon) and the aorta (left colon), described as central vascular ligation. Complete mesocolic excision has been shown to lead to increased lymph node harvest and more mesocolic tissue.

In a comparison between the Leeds and Erlangen units, it was shown that complete mesocolic excision led to an almost doubling in both the number of lymph nodes retrieved and area of mesentery resected. However, a Danish study showed only a 9% increase in lymph node yield.

Surgical concept of complete mesocolic excision represents sharp separation of the undamaged visceral fascia of mesocolon from parietal fascia of peritoneum and the end goal is mobilization of mesocolon and the approach to the appropriate vascular bundle. The scope of surgical intervention depends on localization of the tumor itself. In case that the tumor is located in the right colon next to caecum and ascending colon, it also implies the elevation of duodenum and the head of pancreas (Kocher maneuver) and access to the upper mesenteric vein and artery and its branches. For tumors of the left colon, mobilization of sigma and descending colon is necessary, total separation from the parietal peritoneum, urethra, testicular or ovarian blood vessels, as well as separation from the kidney fat tissue.

The apparent improved outcomes with complete mesocolic excision are yet to be confirmed with a formal Randomized Controlled Trial (RCT). Proposed explanations for the apparent improvements are that increasing lymph node yield permits stage migration, that increased lymph node yield removes a source of metastases, and that it has nothing to do with lymphatics but is due to the preservation of an intact peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven adenocarcinoma (including mucinous and signet-ring cell) or adenosquamous carcinoma on endoscopic biopsy.
* Tumor localization at the caecum, ascending colon, transverse colon, descending colon, sigmoid colon or rectosigmoid on preoperative endoscopy and radiographic imaging [barium enema or computed tomography (CT)] without location of the lower border of the tumor at the rectum.
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.
* Body mass index ≤ 35.
* Sufficient organ function including cardiovascular system and liver.
* Written informed consent.

Exclusion Criteria:

* Contraindications to major surgery and American Society of Anesthesiologists (ASA) Physical Status scoring 4 which means extreme systemic disorders which have already become an eminent threat to life regardless of the type of treatment.
* Infectious disease requiring treatment.
* Body temperature ≥ 38 °C.
* Pregnant women.
* History of psychiatric disease.
* Use of systemic steroids.
* History of myocardial infarction or unstable angina pectoris within 6 months.
* Severe pulmonary emphysema or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Lymph nodes harvest | Day of surgery
  Number of retrieved lymph nodes

SECONDARY OUTCOMES:
Oncologic outcome | 2 years
  Number of patients with local or distant recurrence after the surgery.
Operative outcome | Day of suregry
  A composite outcome of the Operative time, blood loss, blood transfusion, intraoperative morbidities and mortality
Postoperative outcome | 1 month
  A composite outcome of the number of morbidities and mortalities in the postoperative setting
Survival outcome | 3 Years
  Number of patients with 2 year free survival

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelkhalek, M.Sc, Principal Investigator — Oncology Center Mansoura University (OCMU), Egypt; Giovanni Romano, MD, Principal Investigator — National Cancer Institute "Fond. G. Pascale", Italy; Adel Denewer, MD, Study Chair — Oncology Center Mansoura University (OCMU), Egypt; Tamer F Youssef, MD, Study Director — Oncology Center Mansoura University (OCMU), Egypt
Locations (2):
- Oncology Center Mansoura University (OCMU), Egypt, Al Mansurah, Dakahlia Governorate, Egypt
- National Cancer Institute "Fond. G. Pascale", Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817
- [Background] Bertelsen CA, Neuenschwander AU, Jansen JE, Wilhelmsen M, Kirkegaard-Klitbo A, Tenma JR, Bols B, Ingeholm P, Rasmussen LA, Jepsen LV, Iversen ER, Kristensen B, Gogenur I; Danish Colorectal Cancer Group. Disease-free survival after complete mesocolic excision compared with conventional colon cancer surgery: a retrospective, population-based study. Lancet Oncol. 2015 Feb;16(2):161-8. doi: 10.1016/S1470-2045(14)71168-4. Epub 2014 Dec 31. PMID 25555421